CLINICAL TRIAL: NCT06037967
Title: Biobanking for Biomarkers In Respiratory Disease, Allergic Diseases and/or Mast Cell Disorders
Acronym: BIRD-A
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/23/0173
Record Dates: First submitted 2023-09-07; First posted 2023-09-14 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Allergic Diseases; Asthma; Mast Cell Disorders
Keywords: Allergy; asthma; mast cell disorders; biomarkers; biobank
MeSH Terms: conditions — Asthma; Hypersensitivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood sample and tumor tissues
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to build up a clinico-biological bank of samples from patients suspected of or suffering from allergic diseases (including asthma) or mast cell diseases in order to support future research in the field of allergic diseases. The biobank will help to identify new prognostic, diagnostic and/or predictive biomarkers.

DETAILED DESCRIPTION:
This is a prospective monocentric collection of biological samples combined with clinical and paraclinical data from patients suffering from allergic diseases, asthma or mast cell disorders. The aim of this collection is to collect biological samples and clinical data to be used for various exploratory, diagnostic and/or prospective and/or predictive studies.

The samples and data will be pseudonymised, i.e. identified by the first letter of the patient's surname and first name and by a number allocated in chronological order of patient inclusion, and will be stored in a bank. The samples and data making up this clinico-biological bank will be used for subsequent exploratory work used as a priority to answer questions from the Toulouse University Hospital teams in the field of allergic diseases, asthma and/or mast cell disorders, in accordance with the information given to the patient. They may also be transferred to specialised research teams as part of national or international collaborations, or sold to academic or industrial partners. These transfers as part of collaborations or assignments will be legally governed by contracts guaranteeing compliance with the RGPD, where applicable, and the use of these samples in accordance with current legislation and the information provided to patients.

ELIGIBILITY:
Inclusion Criteria:

* patients with a positive prick test or specific IgE regardless of the allergen
* patients suspected of allergic pathology defined by the need to carry out a prick test or specific IgE or a food or drug reintroduction test as part of the treatment
* patients with systemic or cutaneous mastocytosis according to the international classification8
* patients with mast cell activation syndrome according to the international classification8
* patients with familial hyper-alpha tryptasemia on the presence of variation in the number of copies of the alpha allele of the TPSAB1 gene
* patients with asthma of any severity
* people affiliated or beneficiaries of a social security scheme
* patients able to receive and understand the information on the study and their participation and having freely consented to it in writing before any collection of samples or data necessary for the research (no restriction of rights by the judicial authorities and mastery of the French language).

Exclusion Criteria:

* patients under legal protection, guardianship or curatorship
* pregnant or breastfeeding women

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with respiratory disease or allergic disease or mast cell disorders
Sampling Method: Non-Probability Sample
Enrollment: 3200 (Estimated)
Dates: Start 2024-02-28 (Actual); Primary Completion 2038-05 (Estimated); Study Completion 2038-06 (Estimated)

PRIMARY OUTCOMES:
Biobanking for Biomarkers In Respiratory Disease, Allergic diseases and/or mast cell disorders | 15 years
  constitution of a clinico-biological biobanking

SECONDARY OUTCOMES:
set of diagnostic and/or prognostic biomarkers | 15 years
  identify new set of diagnostic and/or prognostic biomarkers
set of predictive biomarkers | 15 years
  Identify new biomarkers and/or a set of predictive biomarkers of the severity of the pathology or the response to treatments.
Allergy markers exploration | 15 years
  Explore if allergy markers (including asthma) or mastocytosis can be found in samples other than blood (urine, skin, etc.).
Estimation of concordance of biomarkers | 15 years
  Estimate the concordance of the presence of known and/or newly identified biomarkers of interest in the biological sample(s) making up the clinical-biological bank with the clinical data collected.
Evolution of biomarkers | 15 years
  Study the evolution over time of the biomarkers of interest and/or newly identified in the biological sample(s) constituting the clinical-biological bank.
Exploration of biological mechanisms | 15 years
  Explore through molecular and/or genomic and/or transcriptomic and/or proteomic studies the biological mechanisms specific to patients with allergic (including asthma) or mast cell pathologies to improve screening, diagnosis, orientation treatment and/or knowledge and understanding of these pathologies

CONTACTS AND LOCATIONS:
Overall Officials: Laurent GUILLEMINAULT, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- Laurent GUILLEMINAULT, Toulouse, France